CLINICAL TRIAL: NCT00548054
Title: Safety and Immunogenicity of a Killed Oral Cholera Vaccine Among Infants 10 Weeks to Less Than 12 Months of Age When Given Concomitantly With EPI Vaccines
Brief Title: Safety and Immunogenicity of a Killed Oral Cholera Vaccine in Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Vaccine Institute (Other)
Collaborators: Indian Council of Medical Research (Other Government); National Institute of Cholera and Enteric Diseases, India (Other); Shantha Biotechnics Limited (Industry); Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CH-WC-01
Record Dates: First submitted 2007-10-21; First posted 2007-10-23 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Cholera; Diarrhea; Vibrio Infections
Keywords: cholera; vaccine; Kolkata; West Bengal; India; immunogenicity; safety; infants; expanded programme on immunization
MeSH Terms: conditions — Cholera; Diarrhea; Vibrio Infections | interventions — shanchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Vaccine Group for Vibriocidal Assay (Experimental): Killed whole cell cholera vaccine bled at day 42 for vibriocidal assay
  Interventions: Biological: Bivalent killed oral cholera vaccine
- Vaccine Group for EPI Assay (Experimental): Killed whole cell cholera vaccine bled at day 56 for EPI immunogenicity testing
  Interventions: Biological: Bivalent killed oral cholera vaccine
- Placebo Group for Vibriocidal Assay (Placebo Comparator): Placebo bled at day 42 for vibriocidal assay
  Interventions: Biological: Killed Escherichia coli K12 placebo
- Placebo Group for EPI Assay (Placebo Comparator): Placebo bled at day 56 for EPI immunogenicity testing
  Interventions: Biological: Killed Escherichia coli K12 placebo
- Vaccine Group for Vibriocidal and Measles Assay (Experimental): Killed whole cell cholera vaccine bled at day 14 and 28 for measles immunogenicity testing
  Interventions: Biological: Bivalent killed oral cholera vaccine
- Placebo Group for Vibriocidal and Measles Assay (Placebo Comparator): Placebo bled at day 14 and 28 for measles immunogenicity testing
  Interventions: Biological: Killed Escherichia coli K12 placebo

INTERVENTIONS:
Biological: Bivalent killed oral cholera vaccine — Oral, 1.5 ml, given 2 times at least 14 days apart
  Other Names: Shanchol
  Arms: Vaccine Group for EPI Assay; Vaccine Group for Vibriocidal Assay; Vaccine Group for Vibriocidal and Measles Assay
Biological: Killed Escherichia coli K12 placebo — oral, 1.5 ml per dose
  Arms: Placebo Group for EPI Assay; Placebo Group for Vibriocidal Assay; Placebo Group for Vibriocidal and Measles Assay

SUMMARY:
In order to assess whether the bivalent killed oral cholera vaccine may be used safely among infants who are most at risk for cholera, the investigators need to determine the safety and immunogenicity of the killed oral cholera vaccine among infants less than 1 year of age when given with the expanded program on immunization (EPI) vaccines including diptheria, pertussis and tetanus (DPT), oral polio vaccine (OPV), Hepatitis B vaccines and measles vaccine. Furthermore, the investigators also need to make sure that immune interference does not occur among all the other vaccine antigens given at the same time. Findings from this study will pave the way for the possible use of the killed whole cell oral cholera vaccine (OCV).

DETAILED DESCRIPTION:
Cholera is an important public health problem worldwide, remaining endemic in most of the developing world at the same time causing outbreaks in areas where lapses in sanitation occur.

A monovalent (anti-O1) oral killed cholera vaccine with a B-subunit was developed by Professor Jan Holmgren in Sweden and is now licensed to a pharmaceutical company in the United Kingdom. The technology for this vaccine was transferred to Vietnamese scientists at the National Institute of Hygiene and Epidemiology in Hanoi in the mid-1980s.

The Vietnamese developed a bivalent vaccine, with killed 0139 cells and without the B-subunit. Since licensure, more than 9 million doses have been given without any report of serious adverse events.

The vaccine has been reformulated in order to internationalize the vaccine. Phase II trials of this vaccine in Son La, Vietnam and Kolkata, India have found the vaccine to be safe with no serious adverse reactions associated with the vaccine. A phase III study of the reformulated vaccine is ongoing in Kolkata, India.

The youngest person the vaccine has been administered to was a 1 year old. Previous studies with the B-subunit containing killed whole cell vaccine was found to be safe among infants as young as 6 months eliciting significant vibriocidal responses among 53% of vaccinees. However, no data is available regarding the use of the bivalent whole cell killed oral vaccine in infants.

Due to the higher risk of cholera among infants, the possibility of introducing cholera vaccine as part of the expanded programme on immunization (EPI) needs to be investigated.

Data regarding the safety and immunogenicity of the reformulated bivalent killed whole cell vaccine among infants needs to be gathered in order to pave the way for the possible use of this vaccine in cholera-endemic areas where infants and children are most at risk. Furthermore, there is no data regarding the concomitant use of this vaccine with other EPI vaccines given to young infants such as Diphtheria-Tetanus-whole cell Pertussis (DTwP), Oral Polio Vaccine (OPV) Hepatitis B and Measles vaccines. It would be important to determine if interference exists between the killed whole cell vaccine and other antigens included in the regular EPI schedule. Providing the killed whole cell vaccine in the context of the EPI will make it easier to introduce cholera vaccines in areas which are cholera-endemic.

ELIGIBILITY:
Inclusion Criteria, Infants 10 weeks to 6 months of age at Day 0:

* Healthy infants aged from birth to 2 months who have not received OPV1, DTP1 or HepB2 will be recruited in Kolkata, North 24 Parganas, and South 24 Parganas
* All subjects must satisfy the following criteria at study entry:

  1. Male or female infants aged from birth to 2 months who the investigator believes will comply with the requirements of the protocol (i.e., available for follow-up visits and specimen collection)
  2. Written informed consent obtained from their parents/guardians
  3. Healthy subjects as determined by:

     * Medical history
     * Physical examination
     * Clinical judgment of the investigator

Inclusion Criteria, Infants 9 months to less than 12 months

* Healthy infants aged from 9 months to less than 12 months who have not received measles vaccine will be recruited in Kolkata, North 24 Parganas, and South 24 Parganas
* All subjects must satisfy the following criteria at study entry:

  1. Male or female infants aged from 9 months to less than 12 months who the investigator believes will comply with the requirements of the protocol (i.e., available for follow-up visits and specimen collection)
  2. Written informed consent obtained from their parents/guardians
  3. Healthy subjects as determined by:

     * Medical history
     * Physical examination
     * Clinical judgment of the investigator

Exclusion Criteria, Infants 10 weeks to 6 months of age at Day 0:

1. Ongoing serious chronic disease
2. Immunocompromising condition or therapy
3. Diarrhea (having more frequent watery stools than usual within a 24 hour period) 6 weeks prior to enrollment
4. Intake of any anti-diarrheal medicine in the past week
5. Irritability, loss of appetite, general ill-feeling or vomiting in the past 24 hours
6. Acute disease one week prior to enrollment, with or without fever. Temperature =>38C (oral) or axillary temperature =>37.5C warrants deferral of the vaccination pending recovery of the subject
7. Receipt of antibiotics in past 14 days
8. Receipt of killed oral cholera vaccine
9. Receipt of live or killed enteric vaccine in 2 months
10. Receipt of DTwP1, OPV1 or Hepatitis B2 vaccines
11. One or two episodes of diarrhea lasting for more than 2 weeks in the past 2 months
12. One or two episodes of abdominal pain lasting for more than 2 weeks in the past 2 months
13. Z-score of < -2 on the weight for age WHO Child Growth Standards

Exclusion Criteria, Infants 9 months to less than 12 months:

1. Ongoing serious chronic disease
2. Immunocompromising condition or therapy
3. Diarrhea (3 or more loose/watery stools within a 24 hour period) 6 weeks prior to enrollment
4. Intake of any anti-diarrheal medicine in the past week
5. Abdominal pain/cramps, loss of appetite, general ill-feeling or vomiting in the past 24 hours
6. Acute disease one week prior to enrollment, with or without fever. Temperature =>38C (oral) or axillary temperature =>37.5C warrants deferral of the vaccination pending recovery of the subject
7. Receipt of antibiotics in past 14 days
8. Receipt of killed oral cholera vaccine
9. Receipt of live or killed enteric vaccine in last 4 weeks
10. Receipt of measles-containing vaccine (MCV)
11. One or two episodes of diarrhea lasting for more than 2 weeks in the past 6 months
12. One or two episodes of abdominal pain lasting for more than 2 weeks in the past 6 months
13. Disease episode potentially related to measles
14. receipt of blood, blood products or a parenteral immunoglobulin preparation in past 3 months
15. History of anaphylaxis, any serious vaccine reaction, allergy to eggs, egg products or to any measles vaccine component
16. Any condition which in the opinion of the investigator might interfere with the evaluation of the study objectives
17. Z-score of < -2 on the weight for age WHO Child Growth Standards

Ages: 10 Weeks to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety: proportion of subjects with diarrhea | entire study period
Immunogenicity: proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies, relative to baseline | 14 days after each dose

SECONDARY OUTCOMES:
Geometric mean serum vibriocidal titers | 14 days after each dose
Proportion of subjects with any of the following: a) immediate reactions 30 minutes and up to 3 days after each dose, b) serious adverse events occurring during the trial, c) any adverse event | entire study period
Proportion of subjects with ≥ 0.1 mIU/ml of anti-diphtheria toxoid antibodies | 28 days after the third DPT dose
Proportion of subjects with ≥ 0.1 mIU/ml of anti-tetanus toxoid antibodies | 28 days after the third DPT dose
For initially seronegative subjects: proportion of subjects with ≥ 15 EU/ml of anti-pertussis IgG and for initially seropositive subjects, proportion with antibody titers equal to or greater than the initial titers prior to vaccination | 28 days after DPT dose
Proportion of subjects with ≥ 10 mIU/ml of anti-HbS antibody | 28 days after the third dose of Hepatitis B vaccine
Proportion of subjects with ≥ 8 fold dilution of anti-polio virus 1, 2, or 3 antibodies by micro-neutralization test | 28 days after the fourth dose of OPV
Proportion of subjects with >150 mIU/ml measles IgG antibodies | 28 days after single dose of measles vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Alok K Deb, PhD, MDDS, Principal Investigator — National Institute of Cholera and Enteric Disease
Locations (1):
- National Institute of Cholera and Enteric Disease, Kolkata, West Bengal, India